CLINICAL TRIAL: NCT04667767
Title: TISA (Traitement Intégré de la Sous-Nutrition Aiguë) Trial : A Cluster Randomized Controlled Trial for the Effect of a WASH Kit Combined With Standard Outpatient Treatment on Severe Acute Malnutrition Recovery in Senegal
Brief Title: The TISA Trial - Senegal
Acronym: TISA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Action Contre la Faim (Other); Cheikh Anta Diop University, Senegal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-KEP-267
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Severe Acute Malnutrition
MeSH Terms: conditions — Severe Acute Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In addition to the national standard outpatient treatment for uncomplicated severe acute malnutrition, caregivers of participants will receive a "WASH kit" containing a plastic container, a supply of Aquatabs® (effervescent chlorine tablets), and training in their use and associated hygiene practices.
  Interventions: Other: WASH kit
- Control (Active Comparator): National standard outpatient treatment for uncomplicated severe acute malnutrition
  Interventions: Other: Standard treatment

INTERVENTIONS:
Other: WASH kit — WASH kit containing a plastic container and a supply of Aquatabs® (effervescent chlorine tablets) and training in their use and associated hygiene practices.
  Arms: Intervention
Other: Standard treatment — National standard outpatient treatment for uncomplicated severe acute malnutrition
  Arms: Control

SUMMARY:
This study evaluates the addition of a simple, scalable "WASH kit", including household water treatment products, a safe water storage container, and hygiene promotion, to the standard national protocol for outpatient treatment of uncomplicated severe acute malnutrition among children aged 6-59 months of age in northern Senegal.

DETAILED DESCRIPTION:
Severe acute malnutrition (SAM) is defined as a weight-for-height z-score (WHZ) below -3 of the World Health Organisation growth standards. It is a short-term acute condition with a high case-fatality rate that increases both the susceptibility of children to infection and the risk of mortality. The global prevalence of SAM in children is estimated to be over 17 million with most of those affected living in sub-Saharan Africa and Asia.

Community-Based Management of Acute Malnutrition (CMAM) has significantly changed standard practice for the treatment of SAM. Uncomplicated SAM cases are now predominantly managed on an outpatient basis and Action Contre la Faim (ACF) supports outpatient treatment programs (OTP) across the globe, particularly in Africa and Asia. This innovation has increased coverage, and reduced the cost of treatment for both the health system and individuals. However, under CMAM, the treatment context has moved from a more controlled health facility setting to the generally less controlled household setting where the risk of infection due to environmental hazards, such as contaminated water, may be higher.

The TISA trial described here will evaluate the effectiveness of combining a simple, scalable "WASH kit" with OTP on the recovery rate among uncomplicated SAM cases aged 6-59 compared to the national standard OTP. The WASH kit includes a plastic container, a supply of Aquatabs® (effervescent chlorine tablets), and training in their use and associated hygiene practices. The study is a cluster randomized controlled trial (cRCT), with health centres constituting the clusters. Clusters are randomly allocated to either a control group receiving the standard OTP or an intervention group receiving OTP plus the WASH kit. The primary outcome of the trial is the recovery rate and the secondary outcomes are weight gain, referral rate, longitudinal prevalence of diarrhoea, prevalence of enteric pathogen detection and all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* Weight-for-height z-score <-3; or
* Brachial perimeter (mid-upper arm circumference) <115; or
* Bilateral oedema

Exclusion Criteria:

* Not able and/or willing to participate for up to 8-weeks
* Clinical complications requiring referral and/or inpatient treatment

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2411 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Rate of recovery | 8 weeks
  Recovery defined as two consecutive weeks with weight-for-height z-scores ≥ -1.5, if admitted based on weight-for-height z-score, or brachial perimeter (mid-upper arm circumference) ≥ 125 mm, if admitted based on brachial perimeter, and no oedema.

SECONDARY OUTCOMES:
Weight gain | 8 weeks
  Weight gain defined as grams of weight gained per kilogram per day between entry and exit.
Rate of referral | 8 weeks
  Referral rate defined as number of participants referred/transferred to next level of care.
Longitudinal prevalence of diarrhoea | 8 weeks
  Longitudinal prevalence is defined by weeks with diarrhoea during follow-up with diarrhoea defined according to WHO definition (3 or more loose or liquid stools passed within 24 hours).
Prevalence of enteric pathogen detection | 8 weeks
  Enteric pathogen detection by stool-based molecular assays of following pathogens: Adenovirus F(40/41), Astrovirus, Norovirus GI, Norovirus GII, Rotavirus, Sapovirus, Enteroaggregative E. coli (EAEC), Shiga-like toxin producing E. coli (STEC), Enteropathogenic Escherichia coli (EPEC), Enterotoxigenic E. coli (ETEC), Shigella/ Enteroinvasive Escherichia coli (EIEC), Campylobacter jejuni/coli, Salmonella enterica, Salmonella enterica Typhi, Vibrio cholerae, Clostridioides difficile, Yersinia enterocolitica, E. coli O157, Aeromonas, Helicobacter pylori, Cryptosporidium spp., Giardia spp., Entamoeba histolytica, Ascaris lumbricoides, Trichuris trichiura, Ancylostoma duodenale, Necator americanus, Strongyloides stercolaris, Plesiomonas shigelloides, Shigella flexneri, Shigella sonnei, Cyclospora cayetanensis.
All cause mortality | 8 weeks
  Deaths occurring during follow-up due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Cumming, MSc, Principal Investigator — London School of Hygiene and Tropical Medicine; Dieynaba N'Diaye, PhD, Principal Investigator — Action Contre La Faim - France; Moustapha Seye, PhD, Principal Investigator — Université Cheikh Anta Diop de Dakar
Locations (1):
- ACF Senegal, Louga, Senegal

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: December 2022
Access Criteria: All IPD that underlie results will be made publicly available

REFERENCES:
- [Derived] N'Diaye DS, Frison S, Ba M, Le ML, Cabo AE, Siroma F, Devort A, MacLeod C, Lapegue J, Seye M, Traore AB, Cerveau T, Leger D, Gallandat K, Gnokane Y, Brizuela AV, Stern S, Braun L, Cumming O. Implementing a pragmatic randomised controlled trial in a humanitarian setting: lessons learned from the TISA trial. Trials. 2024 Sep 19;25(1):620. doi: 10.1186/s13063-024-08459-1. PMID 39300465